CLINICAL TRIAL: NCT05602844
Title: Randomised Controlled Trial Comparing the Outcome of the 3D-Printed Patient-Specific-Instrument Assisted Lapidus Fusion vs Conventional Lapidus Fusion for Surgical Correction of Hallux Valgus Deformity
Brief Title: Clinical Trial on Patient-Specific-Instrumentation Assisted Lapidus Fusion for Hallux Valgus
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Samuel KK Ling, Clinical Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HV PSI Lapidus
Record Dates: First submitted 2022-10-28; First posted 2022-11-02 (Actual); Last update posted 2023-09-25 (Actual); Status verified 2023-09

CONDITIONS: Hallux Valgus; Bunion; Patient Spe
MeSH Terms: conditions — Hallux Valgus; Bunion

STUDY DESIGN:
Intervention Model Description: single-blinded, parallel-group, randomised controlled trial will be conducted to compare the outcome of the 3D-Printed PSI Assisted Lapidus Fusion (n=27) vs Conventional Lapidus Fusion (n=27) for Surgical Correction of HV Deformity
Who Masked: Participant, Outcomes Assessor
Masking Description: Outcome assessment will be performed by orthopaedic surgeons from the Foot and Ankle team; the patient and the outcome assessor will be blinded while the surgeon will not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PSI Lapidus (Experimental): Design of PSI, 3D printing of PSI, PSI-assisted Lapidus Surgery.
  Interventions: Procedure: PSI Lapidus
- Conventional Lapidus (Active Comparator): Lapidus Surgery: exposure of the 1TMTJ via a 3-5cm medial longitudinal skin incision and capsulotomy. Freehand creation of the fusion surface with fluoroscopic assistance. Fixation of the Lapidus arthrodesis will be performed with two 3.5mm headless compression screws.
  Interventions: Procedure: Conventional Lapidus

INTERVENTIONS:
Procedure: PSI Lapidus — Design of PSI: DICOM files will be imported into the Model Intestinal Microflora in Computer Simulation (MIMICS 21.0) 3D image processing software (Materialize, Belgium) for 3D rendering. The segmented bone images will be used for design of the computer-aided modelling (CAM) surgical jigs. 3D printing of PSI jig. PSI-assisted Lapidus Surgery.
  Arms: PSI Lapidus
Procedure: Conventional Lapidus — exposure of the 1TMTJ via a 3-5cm medial longitudinal skin incision and capsulotomy. Freehand creation of the fusion surface with fluoroscopic assistance. Fixation of the Lapidus arthrodesis will be performed with two 3.5mm headless compression screws
  Arms: Conventional Lapidus

SUMMARY:
RCT to compare the effectiveness of PSI assisted Lapidus surgery vs conventional Lapidus surgery in hallux valgus.

DETAILED DESCRIPTION:
Hallux valgus (HV) affects up to 30% of the population. Lapidus surgery, a combination of 1st tarsal-metatarsal joint arthrodesis is one of the most common surgical options for HV. Despite its popularity, the current method alone is not without complications. This will be the world's first Lapidus arthrodesis surgery utilising patient-specific instruments (PSI) as an assistive tool. We hypothesise that PSI will enhance surgical precision, accelerate fusion rates, decrease non-unions, and reduce the need to use bone grafts.

Methods and analysis:

This is a single-blinded, parallel-group, randomised controlled trial comparing the outcome of the 3D-Printed PSI Assisted Lapidus Fusion (n=27) vs Conventional Lapidus Fusion (n=27) for HV deformity. Both groups will receive indentical post-operative rehabilitation of protected weight bearing and splinting. Outcomes measured will include foot function scores, radiological alignment and arthrodesis site assessment with X-ray and High-Resolution Peripheral Quantitative-Computed Tomography, and foot pressure analysis.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic Hallux Valgus
* hallux valgus angle >20
* 1,2 Inter-metatarsal angle >9

Exclusion Criteria:

Individuals with (1) disabilities (both physical and mental) which may impair the adherence of the rehabilitation, (2) revision HV surgery, (3) concomitantly undergone additional procedures on the same foot (e.g. claw toe surgery), (4) the use of medications that may influence bone turnover (e.g. chemotherapy, osteoporotic medications) in recent 3 months, (5) medical comorbidity leading to contraindication for surgery, (6) the inability to understand written Chinese/English, (7) who are mentally/physically unable to consent will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Foot Function | 0 week
  The Foot and Ankle Outcome Score (FAOS) is a reliable and validated patient-reported questionnaire widely used in clinical settings. It consists of five subscales: pain, symptoms, activities of daily living, ability to perform sports and recreational activities, and quality of life. The score of each part is re-coded into a 0-100 scale, with 100 representing no symptoms. (16) The FAOS is a commonly used outcome assessment tool in hallux valgus trials and is reliable and valid by many researchers.
Foot Function | 12 week
  The Foot and Ankle Outcome Score (FAOS) is a reliable and validated patient-reported questionnaire widely used in clinical settings. It consists of five subscales: pain, symptoms, activities of daily living, ability to perform sports and recreational activities, and quality of life. The score of each part is re-coded into a 0-100 scale, with 100 representing no symptoms. (16) The FAOS is a commonly used outcome assessment tool in hallux valgus trials and is reliable and valid by many researchers.
Foot Function | 26 week
  The Foot and Ankle Outcome Score (FAOS) is a reliable and validated patient-reported questionnaire widely used in clinical settings. It consists of five subscales: pain, symptoms, activities of daily living, ability to perform sports and recreational activities, and quality of life. The score of each part is re-coded into a 0-100 scale, with 100 representing no symptoms. (16) The FAOS is a commonly used outcome assessment tool in hallux valgus trials and is reliable and valid by many researchers.
Foot Function | 52 week
  The Foot and Ankle Outcome Score (FAOS) is a reliable and validated patient-reported questionnaire widely used in clinical settings. It consists of five subscales: pain, symptoms, activities of daily living, ability to perform sports and recreational activities, and quality of life. The score of each part is re-coded into a 0-100 scale, with 100 representing no symptoms. (16) The FAOS is a commonly used outcome assessment tool in hallux valgus trials and is reliable and valid by many researchers.
Time to Radiological Fusion | 2 week
  Dorsal-plantar and lateral X-rays of the foot will be taken to look for evidence of trabeculations crossing the fusion site. A successful union will be declared if trabeculation extends more than one-half the length of the fusion site.
Time to Radiological Fusion | 6 week
  Dorsal-plantar and lateral X-rays of the foot will be taken to look for evidence of trabeculations crossing the fusion site. A successful union will be declared if trabeculation extends more than one-half the length of the fusion site.
Time to Radiological Fusion | 12 week
  Dorsal-plantar and lateral X-rays of the foot will be taken to look for evidence of trabeculations crossing the fusion site. A successful union will be declared if trabeculation extends more than one-half the length of the fusion site.
Time to Radiological Fusion | 26 week
  Dorsal-plantar and lateral X-rays of the foot will be taken to look for evidence of trabeculations crossing the fusion site. A successful union will be declared if trabeculation extends more than one-half the length of the fusion site.
Time to Radiological Fusion | 52 week
  Dorsal-plantar and lateral X-rays of the foot will be taken to look for evidence of trabeculations crossing the fusion site. A successful union will be declared if trabeculation extends more than one-half the length of the fusion site.
High-resolution peripheral quantitive-Computed Tomography | 6 week
  HR pQCT allows us to visualize the bony micro-architecture at the Lapidus fusion site and is a more accurate assessment of bone growth compared to X-rays. A rectangular region of interest (ROI) will be established at the fusion surface, inner callus, and external callus area. The volumetric changes in bone mineral density (BMD) in each region will be analyzed.

SECONDARY OUTCOMES:
Deformity severity | 0 week
  Radiology can provide an objective outcome measurement, the 1,2 intermetatarsal angle (IMA) and hallux valgus angle (HVA) will be measured using dorsal-planar weight-bearing X-rays of the foot. The IMA is defined by drawing an angle from lines bisecting the 1st metatarsal and 2nd metatarsal shaft. A normal IMA is <9°, while the more severe the deformity, the larger the angle. The HVA is defined by drawing an angle from the bisecting lines of the 1st proximal phalanx shaft and the 1st metatarsal shaft. A normal HVA is <20° with a larger angle signifying a more severe deformity.
Deformity severity | 12 week
  Radiology can provide an objective outcome measurement, the 1,2 intermetatarsal angle (IMA) and hallux valgus angle (HVA) will be measured using dorsal-planar weight-bearing X-rays of the foot. The IMA is defined by drawing an angle from lines bisecting the 1st metatarsal and 2nd metatarsal shaft. A normal IMA is <9°, while the more severe the deformity, the larger the angle. The HVA is defined by drawing an angle from the bisecting lines of the 1st proximal phalanx shaft and the 1st metatarsal shaft. A normal HVA is <20° with a larger angle signifying a more severe deformity.
Deformity severity | 26 week
  Radiology can provide an objective outcome measurement, the 1,2 intermetatarsal angle (IMA) and hallux valgus angle (HVA) will be measured using dorsal-planar weight-bearing X-rays of the foot. The IMA is defined by drawing an angle from lines bisecting the 1st metatarsal and 2nd metatarsal shaft. A normal IMA is <9°, while the more severe the deformity, the larger the angle. The HVA is defined by drawing an angle from the bisecting lines of the 1st proximal phalanx shaft and the 1st metatarsal shaft. A normal HVA is <20° with a larger angle signifying a more severe deformity.
Deformity severity | 52 week
  Radiology can provide an objective outcome measurement, the 1,2 intermetatarsal angle (IMA) and hallux valgus angle (HVA) will be measured using dorsal-planar weight-bearing X-rays of the foot. The IMA is defined by drawing an angle from lines bisecting the 1st metatarsal and 2nd metatarsal shaft. A normal IMA is <9°, while the more severe the deformity, the larger the angle. The HVA is defined by drawing an angle from the bisecting lines of the 1st proximal phalanx shaft and the 1st metatarsal shaft. A normal HVA is <20° with a larger angle signifying a more severe deformity.
Delayed union rate | 12 week
  Delayed union was defined as greater than 50% lucency on either the AP and lateral radiographs or broken hardware at the fusion site 12 weeks post-surgery. If lucency, sclerosis, or lack of trabeculation extended more than one-half the length of the fusion site on either the dorsal-plantar or lateral radiograph, a radiographic delayed-union was declared
Non-union rate | 26 week
  Non-union was defined as greater than 50% lucency on either the AP and lateral radiographs or broken hardware at the fusion site at 26 weeks post-surgery. If lucency, sclerosis, or lack of trabeculation extended more than one-half the length of the fusion site on either the dorsal-plantar or lateral radiograph, a radiographic non-union was declared
Plantar pressure distribution | 0 week
  The Tekscan Matscan (Tekscan Inc., Boston MA) system will be used to measure the plantar pressure at different anatomical regions during the gait cycle
Plantar pressure distribution | 26 week
  The Tekscan Matscan (Tekscan Inc., Boston MA) system will be used to measure the plantar pressure at different anatomical regions during the gait cycle
Plantar pressure distribution | 52 week
  The Tekscan Matscan (Tekscan Inc., Boston MA) system will be used to measure the plantar pressure at different anatomical regions during the gait cycle

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Ling, Principal Investigator — CUHK
Locations (1):
- CUHK, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
Not shared